CLINICAL TRIAL: NCT03308266
Title: Electromyographic Analysis of the Masticatory Muscles in Cleft Lip and Palate Children With Pain-related Temporomandibular Disorders
Brief Title: Electromyographic Analysis of the Masticatory Muscles in Cleft Lip and Palate Children With Temporomandibular Disorders
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Liliana Szyszka-Sommerfeld, DDS, PhD, Pomeranian Medical University Szczecin
Other Study IDs: KB-0012/08/15
Record Dates: First submitted 2017-10-07; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Cleft Lip and Palate; Temporomandibular Disorder
MeSH Terms: conditions — Cleft Lip; Temporomandibular Joint Disorders | interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CLP children with pain-related TMD
  Interventions: Diagnostic Test: electromyography
- CLP children with no TMD
  Interventions: Diagnostic Test: electromyography
- CLP children with painfree TMD
  Interventions: Diagnostic Test: electromyography

INTERVENTIONS:
Diagnostic Test: electromyography

SUMMARY:
The aim of this study was to assess the electrical activity of the temporal and masseter muscles in cleft lip and palate (CLP) children with pain-related temporomandibular disorders (TMD) and in CLP individuals with no TMD by means of surface electromyography (sEMG). Another objective was to determine the diagnostic value of electromyography in identifying CLP patients with temporomandibular disorders. The sample comprised 87 children with CLP and mixed dentition. The children were assessed for the presence of TMD using of the Research Diagnostic Criteria for TMD (RDC/TMD) by a single examiner. A DAB-Bluetooth Instrument (Zebris Medical GmbH, Germany) was used to take electromyographical (EMG) recordings of the temporal and masseter muscles both in the mandibular rest position and during maximum voluntary contraction (MVC).

ELIGIBILITY:
Inclusion Criteria:

* presence of a cleft without a syndrome, a sequence, or karyotype abnormalities
* presence of mixed dentition

Exclusion Criteria:

* the presence of systemic or rheumatologic diseases
* a history of cervical spine or temporomandibular joint (TMJ) surgery, trauma or malformations

Ages: 6 Years to 13 Years | Sex: All
Age Groups: Child
Study Population: The subjects were selected from patients who had been referred to three Cleft Care Centres in Szczecin, Poznań and Wrocław, Poland.
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Electromyographic analysis of the masticatory muscles in cleft lip and palate children with pain-related temporomandibular disorders | For a single subject the whole EMG examination was taken 40 minutes.
  A DAB-Bluetooth Instrument (Zebris Medical GmbH, Germany) was used to take electromyographical (EMG) recordings of the temporal and masseter muscles both in the mandibular rest position and during maximum voluntary contraction (MVC).Disposable, self-adhesive Ag/AgCl bipolar surface electrodes were placed at a fixed inter-electrode distance of 20 mm on the anterior temporal muscles and on the superficial masseter muscles parallel to the muscular fibres. The EMG signals were amplified, digitized and digitally filtered. The EMG results were analysed using the Student's t test and Mann-Whitney U test to determine differences between the mean values of the independent variables.

SECONDARY OUTCOMES:
The diagnostic value of electromyography in identifying cleft lip and palate patients with temporomandibular disorders | For a single subject the whole EMG examination was taken 40 minutes.
  A DAB-Bluetooth Instrument (Zebris Medical GmbH, Germany) was used to take electromyographical (EMG) recordings of the temporal and masseter muscles both in the mandibular rest position and during maximum voluntary contraction (MVC). Disposable, self-adhesive Ag/AgCl bipolar surface electrodes were placed at a fixed inter-electrode distance of 20 mm on the anterior temporal muscles and on the superficial masseter muscles parallel to the muscular fibres. A mathematical analysis of the ROC curve was used to assess the diagnostic efficiency of electromyography in identifying patients withTMD. The results were described by the area under the curve (AUC), the P value and the ROC coordinate curves, i.e. sensitivity and specificity.

CONTACTS AND LOCATIONS:
Locations (1):
- Pomeranian Medical University, Department of Orthodontics, Szczecin, Poland

REFERENCES:
- [Derived] Szyszka-Sommerfeld L, Machoy M, Lipski M, Wozniak K. The Diagnostic Value of Electromyography in Identifying Patients With Pain-Related Temporomandibular Disorders. Front Neurol. 2019 Mar 5;10:180. doi: 10.3389/fneur.2019.00180. eCollection 2019. PMID 30891001